CLINICAL TRIAL: NCT00380640
Title: The Efficacy of Trimethoprim in Wound Healing of Patients With Epidermolysis Bullosa: A Randomized, Double Blinded, Placebo Controlled, Cross-over Pilot Study
Brief Title: The Efficacy of Trimethoprim in Wound Healing of Patients With Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elena Pope, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1000009064
Record Dates: First submitted 2006-09-25; First posted 2006-09-26 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Epidermolysis Bullosa
Keywords: Pediatrics; Epidermolysis Bullosa; Trimethoprim; Wound Healing
MeSH Terms: conditions — Epidermolysis Bullosa | interventions — Trimethoprim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Trimethoprim
- 2 (Experimental)
  Interventions: Drug: Trimethoprim

INTERVENTIONS:
Drug: Trimethoprim — This group will receive the active intervention (trimethoprim) first, followed by the placebo.
  Arms: 1
Drug: Trimethoprim — This group will start the study with placebo, followed by the active intervention (trimethoprim).
  Arms: 2

SUMMARY:
The purpose of this study is to assess the efficacy of trimethoprim in promoting wound healing and decreasing blister formation in patients with Epidermolysis Bullosa.

DETAILED DESCRIPTION:
Epidermolysis Bullosa (EB) comprises a series of hereditary disorders characterized by fragility of the skin and mucous membranes and the tendency of the skin to blister in response to minor friction or trauma. The care of patients with EB is a complex task that has to be carried out by a multi-professional team. In the absence of a cure, the goal of therapy is the prevention and healing of chronic wounds.

In patients with EB, chronic inflammation interferes with proper wound healing. One treatment option is the use of anti-inflammatory antimicrobial agents, such as trimethoprim, to hasten wound healing and decrease blister formation. This treatment may lead to decreased pain and improvement of the quality of life for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients younger than 20 years of age
* Diagnosis of Recessive Dystrophic Epidermis Bullosa (RDEB)or Junctional Epidermis Bullosa (JEB)
* Signed consent/assent form

Exclusion Criteria:

-Previous known allergy or intolerance to trimethoprim

Ages: 1 Day to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Percentage change of area of the wound from visit to visit, estimated from the longest length and width of up to three target chronic wounds | At 2 months, 3 months and 5 months after baseline visit

SECONDARY OUTCOMES:
Total number of blisters at each visit | At 2 months, 3 months and 5 months after baseline visit
Total number of opened areas at each visit | At 2 months, 3 months and 5 months after baseline visit
Qualitative wound score | At 2 months, 3 months and 5 months after baseline visit
Parent/patient/physician perception of improvement, assessed with a visual analog scale at each visit | At 2 months, 3 months and 5 months after baseline visit
Quality of life, assessed by the Children's Dermatology Life Quality Index (CDLQI) and the Cardiff Wound Impact Schedule | At 2 months, 3 months and 5 months after baseline visit
Number of infections that require systemic antibiotics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Pope, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada